CLINICAL TRIAL: NCT04391621
Title: Efficacy of Autologous Adipose Derived Stromal Vascular Fraction in the Treatment of Keloids
Brief Title: Efficacy of Adipose Derived Stromal Vascular Fraction in the Treatment of Keloids
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC REF 2020-086
Record Dates: First submitted 2019-10-08; First posted 2020-05-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Adipose Derived Stem Cells; Keloid
Keywords: Keloids; Adipose stem cells; Stem cells; Scars
MeSH Terms: conditions — Keloid; Cicatrix | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: Parallel group single centre randomised control pilot trial with a 1:1 ratio.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patients, investigators and outcome assessors will be blinded from the treatment allocation groups. The treatment groups will be recorded such that the assessors will be unaware of the treatment allocations that the participants were involved.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adipose Derived Stem Cell(ADSC) arm (Experimental): In this arm, the participant selected keloid will receive a single dose intra-lesional Adipose derived Stem cells infiltration. This will be harvested and infiltrated as the whole cell pellet (stromal vascular fraction) comprising of an estimate total of 9 million ADSCs (range: 8.4-9.72; SD ± 6.6).
  Interventions: Procedure: Autologous Adipose Derived stem cell transplantation
- Triamcinolone Acetanoide (TAC) arm (Active Comparator): This arm will receive a single dose Triamcinolone acetanoide infiltration into the keloid.
  This will be a single dose infiltration of 40mg/cubic centimetres.
  Interventions: Drug: Triamcinolone Acetonide 40Mg/Ml Inj,Susp_#1

INTERVENTIONS:
Procedure: Autologous Adipose Derived stem cell transplantation — Through liposuction, harvested lipoaspirate will be processed in theatre through centrifugation at 1200g, then the sediment will be washed with Phosphate buffered saline and then incubated at 37 degrees celsius in 0.075% Collagenase type 1a for 1 hour. This will then be washed in an equal volume of 10% Fetal Bovine Serum then filtered through a 100 micrometer cell strainer. Red cells lysed using the Red cell lysis buffer will be performed followed by washing in Phosphate buffered Saline and centrifugation and the stromal vascular fraction cell pellet collected and diluted into 5ml normal saline solution for inflitration. This will then be infiltrated into the affected keloid.
  Other Names: Stromal vasular fraction infiltration
  Arms: Adipose Derived Stem Cell(ADSC) arm
Drug: Triamcinolone Acetonide 40Mg/Ml Inj,Susp_#1 — Triamcinolone Acetanoide 40mg/ml suspension will be diluted into 1ml of 0.5% lignocaine solution and infiltrated into the selected keloid.
  Arms: Triamcinolone Acetanoide (TAC) arm

SUMMARY:
Keloids affect upto 16% of Africans causing significant cosmetic, functional and psychosocial distress. Available treatment options are associated with high recurrence and highly variable symptom relief. Autologous adipose derived stem-cells(ADSCs) have been described to have a potential therapeutic benefit in treating keloids. Investigators will compare intra-lesion single dose Autologous Adipose Derived Stem Cells harvested from abdominal fat to Triamcinolone Acetanoide among 15 patients with keloids treated at Mulago National Referral Hospital in Kampala Uganda between September 2020 and August 2021. These patients will be followed up for keloid volume change at three months following treatment.

DETAILED DESCRIPTION:
Background: Keloids are a disorder of wound healing characterized with excessive scar formation affecting upto 16% of Africans. These are often associated with functional and cosmetic disfigurement with resultant psychosocial distress and reduced quality of life.

Available treatment options are associated with high recurrence and highly variable symptom relief. Autologous Adipose Derived Stem cells (ADSCs) have been recognized to have effect on scar remodeling including regression and remission thus becoming a promising alternative novel therapy. Investigators hypothesize that these ADSCs have a comparable efficacy to Triamcinolone Acetanoide (TAC) which is the existing standard of care in sub-Saharan Africa and therefore intend to evaluate the efficacy and acceptability of ADSCs as a therapy in the treatment of keloids. More specifically they shall evaluate the efficacy and acceptability of ADSCs versus TAC in non-surgical treatment of keloids as well as the efficacy of ADSCs to TAC as post-surgical excision adjuvant therapy in preventing recurrence.

Methods: Investigators shall conduct a single center parallel randomized control trial at Mulago National Referral Hospital following the approval of the Research Ethics Committee of SOM-MakCHS.

For the intervention arm, ADSCs will be obtained by processing lipoaspirate obtained from the abdominal fat-pad of the participants. The control arm will receive TAC. Both arms will receive intra-lesional infiltration of either treatments and followed up at 3 months after therapy. The primary outcome will be the scar regression, remission and acceptability. Two-way Repeated Measures Anova will be used to determine the difference in the treatment arms and time. The All Pair Wise Multiple Comparison Procedure (Holm-Sidak method) will be used to determine the specific differences for both time and treatment factors with an alpha gain set at 0.05.

Potential impact: This project promises to introduce Adipose Derived Stem-cells as a readily available alternative or adjuvant to existing therapies for keloids.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a single keloid of 1-2cm3 as these have the highest response to any treatment administered.

Exclusion Criteria:

* Previous intra-lesional steroid injection treatment in the last three months as the effects may still be ongoing
* Insufficient abdominal fat pad(depth) of 3cm
* Confirmed bleeding disorder
* Ongoing systemic illness
* Ulceration or local keloid infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Keloid regression | 3 months
  The Change in the volume of the keloid tissue in cubic centimetres.

SECONDARY OUTCOMES:
The Patient and Observer Scar Assessment Scale(POSAS) | 3 months
  The pre-treatment and post treatment Patient and Observer Scar Assessment Scale (POSAS) score of the participants will be determined. This is a 10 point score in 1 corresponds to a scar equivalent to normal skin while 10 to the worst possible scar quality. The scar is compared to normal skin at a comparable anatomic site whenever possible.

CONTACTS AND LOCATIONS:
Locations (2):
- Uganda (2):
  - Department of Surgery, Makerere University College of Health Sciences, Kampala
  - Kiruddu National Referral Hospital, Kampala

IPD SHARING:
Plan to Share IPD: No
Will share the IPD only on request.

REFERENCES:
- [Result] Shaffer JJ, Taylor SC, Cook-Bolden F. Keloidal scars: a review with a critical look at therapeutic options. J Am Acad Dermatol. 2002 Feb;46(2 Suppl Understanding):S63-97. doi: 10.1067/mjd.2002.120788. PMID 11807470
- [Result] Davidson S, Aziz N, Rashid RM, Khachemoune A. A primary care perspective on keloids. Medscape J Med. 2009;11(1):18. Epub 2009 Jan 20. PMID 19295939
- [Result] Rockwell WB, Cohen IK, Ehrlich HP. Keloids and hypertrophic scars: a comprehensive review. Plast Reconstr Surg. 1989 Nov;84(5):827-37. doi: 10.1097/00006534-198911000-00021. No abstract available. PMID 2682703
- [Result] Wang X, Ma Y, Gao Z, Yang J. Human adipose-derived stem cells inhibit bioactivity of keloid fibroblasts. Stem Cell Res Ther. 2018 Feb 21;9(1):40. doi: 10.1186/s13287-018-0786-4. PMID 29467010
- [Result] Lee G, Hunter-Smith DJ, Rozen WM. Autologous fat grafting in keloids and hypertrophic scars: a review. Scars Burn Heal. 2017 Apr 6;3:2059513117700157. doi: 10.1177/2059513117700157. eCollection 2017 Jan-Dec. PMID 29799555
- [Result] Ramakrishnan VM, Boyd NL. The Adipose Stromal Vascular Fraction as a Complex Cellular Source for Tissue Engineering Applications. Tissue Eng Part B Rev. 2018 Aug;24(4):289-299. doi: 10.1089/ten.TEB.2017.0061. Epub 2017 Apr 13. PMID 28316259
- [Result] Fan D, Xia Q, Wu S, Ye S, Liu L, Wang W, Guo X, Liu Z. Mesenchymal stem cells in the treatment of Cesarean section skin scars: study protocol for a randomized, controlled trial. Trials. 2018 Mar 2;19(1):155. doi: 10.1186/s13063-018-2478-x. PMID 29499740